CLINICAL TRIAL: NCT02813499
Title: Intérêt de la règle CARE Pour Exclure l'hypothèse d'un Syndrome Coronarien Aigu Sans Dosage Biologique - ICARE
Brief Title: Interest of CARE Rule to Exclude the Hypothesis of an Acute Coronary Syndrome Without Bioassay - ICARE
Acronym: ICARE
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: AOI 2015-06
Record Dates: First submitted 2016-06-10; First posted 2016-06-27 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Chest Pain
Keywords: Acute Coronary Syndrome
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CARE Rule: Evaluation of the clinical suspicion of myocardial infarction and calculation of CARE rule.
  Interventions: Other: CARE Rule

INTERVENTIONS:
Other: CARE Rule — Evaluation of the clinical suspicion of myocardial infarction, calculation of CARE rule and troponin assay performed by the practitioner.

SUMMARY:
Acute coronary syndrome (ACS) is a major health problem and its diagnosis remains a challenge for the emergency physician. The management of a suspected ACS is well codified, based on troponin assays, renewed if necessary.

Conversely, the criteria leading to initiate a diagnostic procedure in chest pain to the Emergency department are unclear. The fear is, firstly, to miss a potentially life treating diagnosis and, secondly, exposing many patients to unnecessary examinations. The advent of highly sensitive troponin assays also increases the risk of over-investigation by a larger number of elevations of the biomarker in non-coronary circumstances leading to a prolongation of hospitalization and, possibly, unnecessary treatments and invasive investigations.

CARE rule could help to streamline this first step. It is established by assigning a value from 0 to 2 to the items: Characteristic of pain, Age, Risk factors and ECG. The search for an ACS is not justified if the sum of points is ≤1 (negative rule) and, conversely, a troponin should be performed if the sum is > 1 (positive rule).

Indeed, CARE rule corresponds to the first 4 items of the HEART score (the latter standing for troponin at admission) whose reliability has been demonstrated, a ≤3 income excluding ACS with a risk of false negatives <2%. A negative CARE rule always corresponds to a HEART score ≤3.

Our study aims to confirm the interest of CARE rule to streamline the search for an ACS in chest pain as an observational European multicenter prospective study.

DETAILED DESCRIPTION:
CARE rule was evaluated in a prospective study of routine care on 641 patients among which 9.8% had a Major Adverse Cardiac Event (MACE). 200 patients (31%) had a negative rule and none showed MACE during the 45-day follow-up (0% [0-1.9]). Among these 200 patients, 119 had a standard troponin assay, a single dosage was increased.

The main objective is to demonstrate the reliability of CARE rule to exclude ACS in chest pain, using an observational Franco-Belgian multicenter study in routine care.

If the reliability of CARE rule is confirmed in Emergency departments, it could be evaluated to be used in other circumstances such as in pre-hospital or in private practice for the general practitioner or cardiologist.

In summary, the ICARE study is intended to allow a rationalization of the management of patients with chest pain, limiting the use of unnecessary investigations while ensuring the safety of care.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted to the emergency department or chest pain
* patient admitted in a non-scheduled manner
* non-traumatic chest pain
* no formal diagnosis after frontline examinations

Exclusion Criteria:

* patient with an ECG showing a coronary syndrome ST +
* patient for which a 6-weeks follow-up would be impossible
* patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with non-traumatic chest pain
Sampling Method: Non-Probability Sample
Enrollment: 1453 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The failure rate of the diagnostic strategy will be evaluated by the rate of MACE recorded in the course of the phone call follow-up at 45 days of patient's inclusion in the group of patients with negative CARE rule. | Day 45
  This rate is a composite criterion including myocardial infarction, percutaneaous coronary intervention, coronary artery bypass grafting or sudden death for which a cardiac cause cannot be excluded. The procedure will be considered acceptable if the rate of false negatives among patients with negative CARE rule is less than 1% with an upper limit of the 95% confidence interval lower than 3%.

SECONDARY OUTCOMES:
The failure rate of the HEART score only considering only one dosage of troponin at admission assessed by the proportion of MACE at 45 days in the HEART group ≤3 | Day 45
Number of bioassay which could be saved, measured by the difference between the number of bioassays actually made least the number bioassays requested by the strategy | Day 45
Difference between average times of consultation according to the need for a bioassay based on CARE rule | Day 45

CONTACTS AND LOCATIONS:
Locations (6):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (5):
  - University Hospital Angers, Angers
  - Hospital of Cholet, Cholet
  - SCHOTTE Thibault, Le Mans
  - Hospital of Saint-Malo, St-Malo
  - University Hospital Toulouse, Toulouse

REFERENCES:
- [Derived] Moumneh T, Penaloza A, Cismas A, Charpentier S, Schotte T, Pernet S, Malatest S, Prunier F, Warnant A, Mezdad TH, Gangloff C, Soulat L, Douillet D, Riou J, Roy PM. Evaluation of HEAR score to rule-out major adverse cardiac events without troponin test in patients presenting to the emergency department with chest pain. Eur J Emerg Med. 2021 Aug 1;28(4):292-298. doi: 10.1097/MEJ.0000000000000791. PMID 34187993